CLINICAL TRIAL: NCT05213975
Title: Effect of Kinesio Taping on Acute Pain, Comfort Level and Breastfeeding Behavior After Cesarean Section: A Randomized Controlled Study
Brief Title: Kinesio Taping Application After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Pinar Uzunkaya Oztoprak, Principal Investigator, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Kinesio Taping
Record Dates: First submitted 2021-12-24; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Pain; Breastfeeding; Caesarean Section;Stillbirth
Keywords: kinesio tape; pain; comfort; breastfeeding
MeSH Terms: conditions — Pain; Breast Feeding | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): kinesio taping group
  Interventions: Device: Kinesio tape
- control group (No Intervention): Standard of care

INTERVENTIONS:
Device: Kinesio tape — Kinesio taping
  Arms: intervention group

SUMMARY:
The study was planned in a randomized controlled study design to determine the effect of kinesio taping applied to women who gave birth by cesarean section on acute pain, comfort level and breastfeeding behavior. The study will be carried out at Hacettepe University Adult Hospital. The universe of the research will be women who gave birth by cesarean section at Hacettepe University Hospital during the study. Women who are planned for a cesarean section, meet the inclusion criteria and volunteer, will be informed about the practice and will be included in the sample of the research. There will be two groups assigned by the randomization method in the study. It is planned that 24 women will be formed in one of them, 48 women in total. In addition to routine treatment and care, kinesio taping will be applied to women in the intervention group; the control group will receive only routine treatment and care.

DETAILED DESCRIPTION:
The study was planned in a randomized controlled study design to determine the effect of kinesio taping applied to women who gave birth by cesarean section on acute pain, comfort level and breastfeeding behavior. The study will be carried out at Hacettepe University Adult Hospital. The universe of the research will be women who gave birth by cesarean section at Hacettepe University Adult Hospital during the study. Women who are planned for a cesarean section, meet the inclusion criteria and volunteer, will be informed about the practice and will be included in the sample of the research. There will be two groups assigned by the randomization method in the study. The number of samples to be recruited into the control and intervention groups was determined by a statistician using the G*Power 3.1.9.4 package program, based on studies in Turkish culture and studies evaluating pain and breastfeeding in women who underwent kinesio taping on the abdominal and breast regions, and the sample size was determined by each of the kinesio taping and control groups. It is planned that 24 women will be formed in one of them, 48 women in total. In addition to routine treatment and care, kinesio taping will be applied to women in the intervention group; the control group will receive only routine treatment and care. The data of the research; "Information Form on Descriptive Characteristics", "Breastfeeding Diagnosis and Evaluation Measurement Tool (LATCH)", "Postpartum Breastfeeding Self-Efficacy Scale" and "Postpartum Comfort Scale", "Visual Analog Scale (Postpartum Breastfeeding Self-Efficacy Scale)" VAS)'' will be collected using the "Mother Follow-up Form". In the analysis of data; in qualitative variables according to descriptive statistics (mean, standard deviation, frequency) and normal distribution of data; Chi-square test, Fisher's exact test, numerical variables; Student's t test, Mann Whitney U test, one-way analysis of variance (ANOVA) and Kruskal Wallis Analysis will be used. Before and after repeated measurements, one-way analysis of variance or Wilcoxon t test will be used according to the normal distribution. At the end of the research, it is expected that the kinesio taping applied after the cesarean section will make a positive contribution to reducing the pain level of the mother, increasing the success of breastfeeding and improving the comfort level.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the research,
* Between the ages of 18- 45,
* At term, delivered by cesarean section and transverse incision applied,
* In the postoperative 8th hour (in the first 6 hours after the operation, hypotension and fatigue due to the effect of the surgery and anesthesia, headache, dizziness, nausea, vomiting, low back pain due to dural puncture are frequently observed, mobilization is delayed [postoperative 6. Hour], in order to have numbness in the extremities, to keep women under the influence of anesthesia cognitively, and to perform measurement tools and taping effectively, the application will be started from the 8th postoperative hour.),
* Having a single and healthy baby,
* Do not have a breast problem that prevents milk secretion (such as undergoing breast augmentation/reduction surgery, mass, endocrine disease, etc.),
* Not having nipple problems that may affect breastfeeding (nipple turned inward, flat, numerous and drooping at the size of a bottle head, etc.),
* No history of breast cancer,
* Does not have a dermatological disease,
* No migraine or similar chronic pain,
* Women who do not have intellectual disability or perception problems and do not have communication difficulties will be included in the research.

Exclusion Criteria:

* Having a diagnosis of allergic disease on the skin,
* Developing postpartum complications (bleeding, infection, fever, etc.),
* Women whose babies were taken to the neonatal intensive care unit will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
pain level | 4 months
  Pain level between 0 and 100 will be determined by scoring using the VAS scale.
The Breastfeeding Self-Efficacy Scale | 4 months
  The Breastfeeding Self-Efficacy Scale was first developed by Dennis and Faux (1999) as a 33-item scale. This scale assesses how competent mothers feel about breastfeeding. All items in the scale have positive meaning. The Turkish adaptation of the scale was made by Alush-Tokat and Okumuş (2010). The cronbach's alpha value of the scale was found to be 0.86, and it was found to be a reliable scale. The Breastfeeding Self-Efficacy Scale consists of 14 items assessing breastfeeding self-efficacy. The scale is a 5-point Likert type scale and is evaluated as I am never sure (1 point) and I am always sure (5 points). The minimum score that can be obtained from the scale is 14, and the maximum score is 70. The scale has no cut-off point and an increase in the score means higher breastfeeding self-efficacy (Dennis & Faux, 1999; Dennis, 2003).
Postpartum Comfort Scale | 4 months
  Developed by Karakaplan and Yıldız (2010) in line with the comfort theory developed by Katharine Kolcaba in 1994, the Postpartum Comfort Scale consists of 34 items. The scale can evaluate postpartum comfort in 3 dimensions (physical, psychospiritual, sociocultural). The scale is evaluated using a 5-point Likert-type scale scoring system, ranging from "strongly agree" (5 points), to "strongly disagree" (1 point) for each item. In positive sentences, I completely agree indicates the best comfort (5 points), and negative sentences indicate low comfort (1 point). The total score obtained from the scale is divided by the number of items to determine an average of 18 values, and the result is shown in the 1-5 distribution. Accordingly, the lowest score to be taken from the scale is 34, and the highest score is 170 (Karakaplan & Yildiz, 2010).
Breastfeeding Diagnostic and Evaluation Measurement Tool (LATCH) | 4 months
  The scale was developed by Jensen, Wallace and Kelsay in 1994 by analogy with the APGAR score system. It was created to make the diagnosis of breastfeeding objectively, to determine breastfeeding problems and to make a training plan, to create a common language among healthcare professionals about breastfeeding and to use it in research (Jensen et al., 1994). The Turkish validity of the Measurement Tool was found to be between 0.94 and 0.96 in studies (Demirhan, 1997; Küçükoğlu, 2011).
  For each criterion that makes up the LATCH Breastfeeding Diagnostic and Evaluation Scale, 0, 1, 2 points are given. Breastfeeding success is evaluated by summing the scores. The highest score that can be obtained from the scale is 10 and the lowest score is 0. A score below 10 points for mothers indicates that they need support in breastfeeding, and as the score decreases, mothers' need for breastfeeding support increases (Jensen et al., 1994; Demirhan, 1997; Küçükoğlu, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Ozgür Ozyüncü, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, CSR
Time Frame: january 2023
Access Criteria: Statistical analyzes of the study will be made by an expert. The data will be shared with the expert by providing statistical blinding. The results of the study will be published in an international journal.